CLINICAL TRIAL: NCT07235254
Title: Dry Versus Moist Ag Dressings for Local Wound Infections: A Randomized Controlled Trial on Effectiveness and Cost-Effectiveness
Brief Title: A RCT of Moist Ag Dressing in Chronic Wound
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Long Zhang, Head of Wound Healing Center, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Long2025-CW-Ag foam dressing
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Chronic Wound; Hard to Heal Wounds; Dressing; Wound he'a'Ling; Wound Healing

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOIST Ag dressing (Experimental): Using MepilexAg in conjunction with conventional clinical treatments
  Interventions: Device: Ag foam dressing named MepilexAg
- Dry Ag dressing (Active Comparator): Using dry Ag dressing in conjunction with conventional clinical treatments
  Interventions: Device: Dry Ag dressing

INTERVENTIONS:
Device: Ag foam dressing named MepilexAg — Using MepilexAg in conjunction with conventional clinical treatments in chronic local infectious ulcer
  Arms: MOIST Ag dressing
Device: Dry Ag dressing — Using dry Ag dressing in conjunction with conventional clinical treatments
  Arms: Dry Ag dressing

SUMMARY:
This study aims to explore the differences in efficacy and cost-effectiveness between self-adhesive soft polysilicone silver ion foam dressings and traditional silver dressings in local infected wounds through a prospective randomized controlled study. The goal is to provide evidence-based medical support for clinical application, further shorten the wound healing time, and reduce the economic burden on the medical system and patients.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's age ranges from 18 to 80 years old.
2. According to the IWII wound infection staging, infected wounds are classified as local infections*.
3. The wound type is ulcer, with an ulcer area ranging from 1 to 40 cm².
4. The wound stage is in the necrosis stabilization phase, granulation growth phase, or epithelial crawling phase**.
5. Voluntary participation in this study and signing the informed consent form

Exclusion Criteria:

1. Severe diseases such as acute myocardial infarction, heart failure, hepatitis, shock, and respiratory failure have not been corrected yet;
2. The blood sugar level of diabetes is out of control, with fasting blood sugar > 15 mmol/L and glycosylated hemoglobin ≥ 10%;
3. There is active bleeding in the wound, and the conventional basic treatment plan cannot be implemented;
4. Serum albumin < 20 g/L; hemoglobin < 60 g/L; platelets < 50 × 109/L;
5. Disseminated infection or systemic infection state, and antibiotics are being used or will be used for treatment;
6. Patients with advanced malignant tumors;
7. The patient is in the active stage of autoimmune diseases;
8. The patient has previously been allergic to self-adhesive soft polysilicone silver ion foam dressings (Meipikang Silver) or Anxidean Nano Silver Trauma Patch;
9. The patient cannot cooperate or has a mental disorder;
10. According to the investigator's judgment, the subject has clear reasons that affect wound healing and is not suitable for this study or cannot comply with the requirements of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
wound area reduction in two weeks | From enrollment to the end of treatment at 2 weeks
  Pre-treatment area minus post-treatment area, then divided by pre-treatment area

SECONDARY OUTCOMES:
wound healing rate | From enrollment to the end of treatment at 2 weeks
  Percentage of healed wounds to total cases by D14

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided